CLINICAL TRIAL: NCT06457061
Title: Evaluation of Caregiver Burden and Depression Severity in Patients With Right and Left Hemiplegia
Brief Title: Evaluation of Caregiver Burden and Depression Severity in Patients With Hemiplegia
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-SK-06
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hemiplegia; Caregiver Burden; Depression
MeSH Terms: conditions — Hemiplegia; Caregiver Burden; Depression | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Right Hemiplegia
  Interventions: Other: Survey Study
- Left Hemiplegia
  Interventions: Other: Survey Study

INTERVENTIONS:
Other: Survey Study — Barthel Index for Activities of Daily Living Scale, Beck Depression Inventory and Star Cancellation Test questionnaires were applied to hemiplegia patients.
  Beck Depression Inventory and Zarit Caregiver Burden Interview surveys were administered to caregivers.

SUMMARY:
This study aimed to evaluate the caregiving burden and severity of depression in patients with right hemiplegia and left hemiplegia.

DETAILED DESCRIPTION:
Stroke is a disease characterized by neurological symptoms and signs lasting more than 24 hours, which can lead to death after the interruption of brain blood flow or due to focal brain damage. Post-stroke disability affects the patient's quality of life, makes the patient dependent on the caregiver, creates a caregiver burden, and brings socioeconomic and social consequences. Different hemispheres of the brain undertake different tasks. Different clinical conditions may occur in stroke patients with right or left hemiplegia following cerebrovascular infarction. This may affect the care burden of caregivers and the severity of depression. It was thought that knowing the care burden of patients with right and left hemiplegia would positively contribute to the quality of care given to patients.This study aimed to evaluate the caregiving burden and severity of depression in patients with right hemiplegia and left hemiplegia.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia patients between the ages of 18 and 75 were included.
* Caregivers over 18 years of age
* At least 3 months must have passed since the patient was diagnosed.
* Caregivers of patients should be their first and second degree relatives.
* Caregivers must be competent to understand what they read and complete the questionnaires.
* Caregivers must have been caring for their patients for at least 3 months.

Exclusion Criteria:

* Patients and caregivers with a history of psychiatric illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemiplegia patients treated in our outpatient and inpatient physical therapy and rehabilitation units and their first- or second-degree relatives who care for these patients constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Beck's Depression Inventory | Day 1
  The Beck Depression Inventory (BDI) is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression. The score to be received varies between 0-63. A high total score indicates a higher severity of depression.
Zarit Caregiver Burden | Day 1
  Zarit caregiver burden interview evaluates caregivers' caregiving burden. It consists of 22 questions. A minimum of 0 and a maximum of 88 points can be obtained from the scale. A A high total score indicates a higher severity of caregiver burden

SECONDARY OUTCOMES:
Barthel Index for Activities of Daily Living Scale | Day 1
  The Barthel index is used to assess activities of daily living. It consists of 10 items: feeding, bathing, grooming, dressing, bowel, bladder, toilet use, transfers, mobility, stairs. Scores range from 0-100. A score of 100 represents complete independence, and a score of 0 represents complete dependence.
Star Cancellation test | Day 1
  The Star Cancellation Test is a screening tool developed to detect the presence of unilateral spatial neglect

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No